CLINICAL TRIAL: NCT05500417
Title: First-in-Human Safety and Immunogenicity Evaluation of an Intramuscular Campylobacter Jejuni Conjugate Vaccine (CJCV2) With and Without Army Liposome Formulation Containing QS-21 (ALFQ)
Brief Title: Safety and Immunogenicity of CJCV2 With and Without ALFQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-0003; 5UM1AI148372-03 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-02-07

CONDITIONS: Campylobacter Infection
Keywords: ALFQ; Campylobacter jejuni; Campylobacter jejuni Conjugate Vaccine; CJCV2; Immunogenicity; QS-21; safety
MeSH Terms: conditions — Campylobacter Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1A (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 1 microgram of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Biological: CJCV2
- Group 1B (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 1 microgram of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) and a full dose of Army Liposome Formulation containing QS-21 (ALFQ) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Drug: ALFQ; Biological: CJCV2
- Group 2A (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 3 micrograms of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Biological: CJCV2
- Group 2B (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 3 micrograms of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) and a full dose of Army Liposome Formulation containing QS-21 (ALFQ) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Drug: ALFQ; Biological: CJCV2
- Group 3A (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 10 micrograms of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Biological: CJCV2
- Group 3B (Experimental): Each subject will receive a 1 mL intramuscular (IM) injection containing 10 micrograms of Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) and a full dose of Army Liposome Formulation containing QS-21 (ALFQ) on Days 1, 29, and 57. 3 sentinel subject will be dosed first; if no safety signals are noted within 7 days after sentinel dosing, the remaining 7 subjects will be dosed. N=10
  Interventions: Drug: ALFQ; Biological: CJCV2

INTERVENTIONS:
Drug: ALFQ — ALFQ (Army Liposome Formulation containing QS-21) is composed of ALF55 (cGMP-manufactured Army Liposome Formulation), QS-21 (purified extracted saponin), and Sorensen's Phosphate Buffer. Full dose of AFLQ compromised of 200 microgram 3D-PHAD and 100 microgram QS-21, co-administered with main intervention.
  Arms: Group 1B; Group 2B; Group 3B
Biological: CJCV2 — Vaccine comprised of C. jejuni capsule conjugated to Cross-Reactive Material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin. CJCV2 will be reconstituted in 1 mL of sterile water for injection (SWI). The resuspended CJCV2 product will be diluted with sterile 0.9% Sodium Chloride for Injection. 3 dosages for administration: 1 microgram, 3 micrograms, and 10 micrograms.

SUMMARY:
This is a randomized, double-blind, dose-escalating, outpatient trial in a total of approximately 60 subjects, assigned to 3 cohorts (20 subjects per cohort). Each subject will receive one of three intramuscular (IM) vaccinations, spaced 28 days apart, of Campylobacter jejuni Conjugate Vaccine (CJCV2) with or without a fixed dose of the adjuvant Army Liposome Formulation containing QS-21 (ALFQ)(200 mcg 3D-PHAD, 100 mcg QS-21). Three doses (1 ug, 3 ug and 10 ug) of CJCV2 will be evaluated. The first six participants at each dose will be sentinels and randomized in a 1:1 blinded fashion to receive CJCV2 with or without ALFQ. The primary objective is to evaluate the safety of the three different doses of IM injection of CJCV2 with and without ALFQ. The study hypothesis is that the CJCV2 vaccine alone and CJCV2 with ALFQ adjuvant will be safe and that the CJCV2 alone will be immunogenic, with immunogenicity enhanced through the use of the adjuvant ALFQ.

DETAILED DESCRIPTION:
This is a randomized, double-blind, dose-escalating, outpatient trial in a total of approximately 60 subjects, assigned to 3 cohorts (20 subjects per cohort). Each subject will receive one of three intramuscular (IM) vaccinations, spaced 28 days apart, of Campylobacter jejuni Conjugate Vaccine (CJCV2) with or without a fixed dose of the adjuvant Army Liposome Formulation containing QS-21 (ALFQ)(200 mcg 3D-PHAD, 100 mcg QS-21).Three doses (1 ug, 3 ug and 10 ug) of CJCV2 will be evaluated. The first six participants at each dose will be sentinels and randomized in a 1:1 blinded fashion to receive CJCV2 with or without ALFQ. The primary objective is to evaluate the safety of the three different doses of IM injection of CJCV2 with and without ALFQ. The secondary objective is to evaluate C. jejuni capsule-specific serum IgG responses following vaccination. The study hypothesis is that the CJCV2 vaccine alone and CJCV2 with ALFQ adjuvant will be safe and that the CJCV2 alone will be immunogenic, with immunogenicity enhanced through the use of the adjuvant ALFQ.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent prior to initiation of any study procedures.
2. Able to understand and comply with planned study procedures and be available for all study visits/safety communications.
3. Non-pregnant/non-lactating subjects 18-50 years of age inclusive upon enrollment.
4. In general, good health* to be safely enrolled in this study as determined by medical history, medication use**, and physical exam.

   *Good health is defined by the absence of any exclusionary medical conditions. If the subject has another current, ongoing medical condition, the condition cannot meet any of the following criteria; 1) first diagnosed within 3 months of enrollment; 2) is worsening in terms of clinical outcome in last 6 months; or 3) involves need for medication that may pose a risk to subject's safety or impede assessment of AEs or immunogenicity if they participate in the study.

   **Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion #17). Herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.4 degrees F.
6. Pulse is 50 to 100 beats per minute (bpm), inclusive.
7. Systolic blood pressure (BP) is 90 to 140 mmHg, inclusive.
8. Diastolic BP is 55 to 90 mmHg, inclusive.
9. Body Mass Index(BMI) less than 40.
10. Females of childbearing potential* may enroll if subject has practiced adequate contraception** > 30 days prior to enrollment and agrees to continue adequate contraception for the entire study.

    *Child-bearing potential is defined as not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

    **Adequate contraception includes; non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide, effective intrauterine devices, NuvaRing (R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
11. Females of childbearing potential must have a negative urine pregnancy test within 24 hours prior to enrollment.
12. Agree not to participate in another interventional clinical trial during the study period that may affect the analysis or endpoint assessment.
13. Negative urine drug screen for opiates.

Exclusion Criteria:

1. Have any disease or medical condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute or chronic disease or medical condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.

   These include:

   History of inflammatory bowel disease (IBD) (including ulcerative colitis, Crohn's disease, indeterminate colitis, or celiac disease). Within the past 12 months, has any of the following: irritable bowel syndrome (IBS) or any active uncontrolled gastrointestinal disorders or diseases as assessed by the investigator, including symptoms or evidence of active gastritis or gastroesophageal reflux disease, gastric surgery or gastric acid hyper-secretory disorders (e.g., Zollinger-Ellison syndrome), gastrointestinal obstruction, ileus, gastric retention, bowel perforation, toxic colitis, persistent infectious gastroenteritis, persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection. History of immunodeficiency due to congenital or hereditary causes, underlying illness or treatment, autoimmune disorders, or chronic inflammatory disorders. History of an inflammatory arthritis such as reactive arthritis, Reiter's syndrome, ankylosing spondylitis, rheumatoid arthritis, or GBS. Known active neoplastic disease non-melanoma, treated, skin cancers are permitted, a history of any hematologic malignancy, or have used anticancer chemotherapy/radiation therapy (cytotoxic) within 5 years prior to study vaccination. Other condition requiring daily therapy that would place the volunteer at increased risk or Adverse Events (AE). Other laboratory abnormalities which in the opinion of the investigator precludes participation in the study. Clinically significant abnormalities on physical exam.
2. Documented history of auto-immune conditions in a first-degree relative. Examples include reactive arthritis, Reiter's syndrome, ankylosing spondylitis, rheumatoid arthritis, or GBS.
3. History of Potentially Immune-Mediated Medical Conditions (PIMMCs).
4. Evidence of inflammatory arthritis on exam and/or positive serology results for HLA-B27.
5. Positive Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C antibodies (HCVs).
6. Participation in a previous Campylobacter study or reports having received vaccination against Campylobacter within the last 3 years.
7. History of microbiologically confirmed Campylobacter infection in the last 3 years.
8. Occupation involving handling of Campylobacter bacteria or vaccine products currently or in the past 3 years.
9. Use of immunosuppressive/immunomodulating disease therapy within 90 days
10. Received Immunoglobulin (Ig) or other blood products (with exception of Rho D Ig) within 90 days prior to enrollment.
11. Have a history of severe reactions following previous immunization with any licensed or unlicensed vaccine.
12. Known hypersensitivity to any components of vaccine, adjuvant or diluent.
13. Received or plan to receive a licensed live vaccine within 30 days prior to 1st vaccination and to 30 days after the last vaccination.
14. Received or plan to receive a licensed, inactivated, vaccine within 14 days prior to 1st vaccination to 14 days after the last vaccination, or a seasonal influenza and/or COVID-19 vaccine +/- 7 days from study product vaccination.
15. Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is unacceptably obscured due to a physical condition or permanent body art.
16. Within 14 days prior to vaccination has received an oral or parenteral (including intra-articular) corticosteroid of any dose for 5 or more days, or high-dose inhaled corticosteroids. a) High dose defined per age as using inhaled high dose per reference chart (https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf)
17. Current or history of alcohol or drug abuse within one year prior to enrollment.
18. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
19. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within one year prior to enrollment.
20. Are pregnant, breastfeeding, or plan to become pregnant or breastfeed at any given time during the study.
21. Have an acute illness as determined by study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site PI or sub-investigator, within 72 hours prior to enrollment.

    a. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site PI or sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
22. Received an investigational product within 30 days prior to the first study vaccination or expect to receive an investigational product during the study period.

    a. Including vaccine, drug, biologic, device, blood product, or medication, other than from participation in this trial.
23. Have abnormal screening laboratory values within 30 days prior to enrollment. a. Screening laboratory values that are outside acceptable range but are thought to be due to an acute condition or due to laboratory error may be repeated once.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was comprised of generally healthy young adults (males and non-pregnant or -lactating females) 18-50 years of age, inclusive, who met all eligibility criteria. Participants were recruited from existing volunteer populations and from the communities at large around the clinical site. Fifty-nine participants were enrolled between 13Sep2022 and 08Nov2023.
Groups:
- 1 µg CJCV2: 1 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
- 1 µg CJCV2 + ALFQ: 1 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
  Army Liposome Formulation containing QS-21 (ALFQ) is a combination adjuvant composed of ALF55, QS-21, and Sorensen's Phosphate Buffer. ALF55 is an Army Liposome Formulation (ALF) containing the phospholipids dimyristoyl phosphatidyl choline and dimyristoyl phosphatidyl glycerol, 3D-PHAD®, and 55% cholesterol. QS-21 is a purified saponin extracted from the bark of the Quillaja saponaria tree. ALFQ was manufactured at the Walter Reed Army Institute for Research (WRAIR) Pilot Bioproduction Facility (Silver Spring, Maryland).
- 3 µg CJCV2: 3 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
- 3 µg CJCV2 + ALFQ: 3 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
  Army Liposome Formulation containing QS-21 (ALFQ) is a combination adjuvant composed of ALF55, QS-21, and Sorensen's Phosphate Buffer. ALF55 is an Army Liposome Formulation (ALF) containing the phospholipids dimyristoyl phosphatidyl choline and dimyristoyl phosphatidyl glycerol, 3D-PHAD®, and 55% cholesterol. QS-21 is a purified saponin extracted from the bark of the Quillaja saponaria tree. ALFQ was manufactured at the Walter Reed Army Institute for Research (WRAIR) Pilot Bioproduction Facility (Silver Spring, Maryland).
- 10 µg CJCV2: 10 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
- 10 µg CJCV2 + ALFQ: 10 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
  Campylobacter jejuni Conjugate Vaccine 2 (CJCV2) is a purified HS23/36 capsular polysaccharide (CPS) of Campylobacter jejuni (C. jejuni) conjugated to cross-reactive material 197 (CRM197), a non-toxic mutant protein of diphtheria toxin, at a CPS:CRM197 ratio of 2:1. The CJCV2 vaccine product was manufactured at Inventprise LLC (Redmond, Washington) with final fill and finish completed by The University of Iowa Pharmaceuticals (Iowa City, Iowa).
  Army Liposome Formulation containing QS-21 (ALFQ) is a combination adjuvant composed of ALF55, QS-21, and Sorensen's Phosphate Buffer. ALF55 is an Army Liposome Formulation (ALF) containing the phospholipids dimyristoyl phosphatidyl choline and dimyristoyl phosphatidyl glycerol, 3D-PHAD®, and 55% cholesterol. QS-21 is a purified saponin extracted from the bark of the Quillaja saponaria tree. ALFQ was manufactured at the Walter Reed Army Institute for Research (WRAIR) Pilot Bioproduction Facility (Silver Spring, Maryland).
Period: Overall Study
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Started | 10 | 10 | 10 | 10 | 9 | 10
Completed | 10 | 10 | 10 | 9 | 9 | 10
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 µg CJCV2: 1 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
- 1 µg CJCV2 + ALFQ: 1 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
- 3 µg CJCV2: 3 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
- 3 µg CJCV2 + ALFQ: 3 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
- 10 µg CJCV2: 10 µg of CJCV2 administered intramuscularly on Days 1, 29, and 57.
- 10 µg CJCV2 + ALFQ: 10 µg of CJCV2 with fixed dose (200 µg 3D-PHAD®, 100 µg QS-21) of ALFQ, administered intramuscularly on Days 1, 29, and 57.
- Total: Total of all reporting groups
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.9) | 31.9 (6.7) | 39.8 (7.2) | 34.4 (9.3) | 38.1 (6.6) | 33.8 (8.2) | 34.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 7 | 5 | 7 | 37
  Male | 5 | 3 | 4 | 3 | 4 | 3 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 8 | 9 | 10 | 9 | 9 | 10 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 0 | 1 | 4
  White | 9 | 7 | 9 | 8 | 8 | 7 | 48
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 10 | 10 | 10 | 10 | 9 | 10 | 59
Height [Mean (Standard Deviation); unit: cm] | 174.44 (13.59) | 171.60 (7.96) | 174.10 (11.24) | 167.05 (10.45) | 175.89 (12.57) | 171.55 (14.19) | 172.38 (11.68)
Weight [Mean (Standard Deviation); unit: kg] | 82.39 (24.76) | 75.21 (14.15) | 87.89 (18.10) | 76.28 (11.70) | 79.81 (18.00) | 84.87 (25.57) | 81.10 (19.11)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.50 (5.13) | 25.68 (5.30) | 29.04 (5.49) | 27.38 (3.74) | 25.83 (5.70) | 28.58 (6.55) | 27.19 (5.30)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Solicited Local Adverse Events (AEs) Through 7 Days After Each Study Vaccination
Description: Solicited local AEs were collected 30 minutes post-vaccination, and then daily for 7 days after each vaccination using a memory aid and graded on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe). Local symptoms included ecchymosis, ecchymosis (measurement), erythema, erythema (measurement), induration/edema, induration/edema (measurement), pain, and tenderness.
Time Frame: Days 1 through 8, Days 29 through 36, and Days 57 through 64
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants
  Post-Vaccination 1 | 4 | 9 | 2 | 10 | 5 | 7
  Post-Vaccination 2: number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9
  Post-Vaccination 2 | 2 | 8 | 3 | 8 | 4 | 9
  Post-Vaccination 3: number analyzed (Participants) | 10 | 10 | 10 | 8 | 9 | 9
  Post-Vaccination 3 | 6 | 8 | 2 | 7 | 3 | 7

2. Primary Outcome: Number and Percentage of Participants With Solicited Systemic Adverse Events (AEs) Through 7 Days After Each Study Vaccination
Description: Solicited systemic AEs were collected prior to vaccination, 30 minutes post-vaccination, and then daily for 7 days after each vaccination using a memory aid and graded on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe). Systemic symptoms included arthralgia, fatigue, fever, feverishness (chills/shivering/sweating), headache, malaise, myalgia, nausea, and vomiting.
Time Frame: Days 1 through 8, Days 29 through 36, and Days 57 through 64
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants
  Post-Vaccination 1 | 7 | 9 | 5 | 9 | 6 | 8
  Post-Vaccination 2: number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9
  Post-Vaccination 2 | 5 | 10 | 4 | 8 | 4 | 7
  Post-Vaccination 3: number analyzed (Participants) | 10 | 10 | 10 | 8 | 9 | 9
  Post-Vaccination 3 | 6 | 9 | 5 | 6 | 3 | 7

3. Primary Outcome: Number and Percentage of Participants With Vaccine-related Unsolicited AEs Through 28 Days Post Last Vaccination
Description: ICH E6 defines an AE as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, regardless of its causal relationship to the study treatment. The FDA defines an AE as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. The occurrence of an AE could have come to the attention of study personnel during study visits and interviews of a study participant presenting for medical care, or upon review by a study monitor.
  An AE was considered related if there was a reasonable possibility that the study product caused the AE. Reasonable possibility means that there was evidence to suggest a causal relationship between the study product and the AE.
Time Frame: Day 1 through Day 85
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants | 1 | 0 | 1 | 2 | 0 | 0

4. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events (SAEs)
Description: An AE or suspected adverse reaction was considered a SAE if, in the view of either the PI or sponsor, it resulted in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not have resulted in these outcomes could be considered serious when, based upon appropriate medical judgment, they could have jeopardized the participant and could have required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 420
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants | 0 | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number and Percentage of Participants With Medically Attended Adverse Events (MAAEs) From First Study Vaccination Through End of Study Participation
Description: Medically attended adverse events (MAAEs) are any unsolicited AE for which a participant received medical attention, defined as hospitalization, an ER visit, or an otherwise unscheduled visit to or from medical personnel.
Time Frame: Day 1 through Day 420
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants | 5 | 3 | 3 | 7 | 5 | 6

6. Primary Outcome: Number and Percentage of Participants With New-onset Chronic Medical Conditions (NOCMCs) From First Study Vaccination Through End of Study Participation
Description: New-onset chronic medical conditions (NOCMCs) are defined as any new ICD-10 diagnosis that is applied to the participant during the duration of the study, after receipt of the study product, that is expected to continue for at least 3 months and requires continued health care intervention.
Time Frame: Day 1 through Day 420
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants | 1 | 0 | 0 | 0 | 1 | 2

7. Primary Outcome: Number and Percentage of Participants With Potentially Immune-mediated Medical Conditions (PIMMCs) From First Study Vaccination Through End of Study Participation
Description: Potentially immune-mediated medical conditions (PIMMCs) constitute a group of AEs that includes diseases which are clearly autoimmune in etiology and other inflammatory and/or neurologic disorders which may or may not have autoimmune etiologies.
Time Frame: Day 1 through Day 420
Population: The Safety Population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With >= 4-fold Rise From Baseline in C. Jejuni Capsule-specific Immunoglobulin G (IgG) Serum Antibodies
Description: Serum from blood collected at Study Days 1, 8, 29, 36, 57, 64, 85, and 113 was analyzed using an enzyme-linked immunosorbent assay (ELISA) to measure C. jejuni capsule-specific Immunoglobulin G (IgG) serum antibody titers. Results below the lower limit of quantification (LLOQ) were imputed as LLOQ/2. The percentage of participants with at least a 4-fold rise in antibody titer compared to pre-vaccination 1 is presented by arm with exact 95% Clopper-Pearson confidence interval.
Time Frame: Days 8, 29, 36, 57, 64, 85, and 113
Population: The Full Immunogenicity Population consists of all participants who received any study product and contributed both pre- and at least one post-study vaccination blood samples for immunogenicity testing for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 10
Percentage of participants
  Day 8 | 0.0 [0.0 to 30.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 3.8]
  Day 29 | 0.0 [0.0 to 30.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 33.6] | 10.0 [0.3 to 44.5]
  Day 36 | 20.0 [2.5 to 55.6] | 70.0 [34.8 to 93.3] | 10.0 [0.3 to 44.5] | 100.0 [66.4 to 100.0] | 33.3 [7.5 to 70.1] | 60.0 [26.2 to 87.8]
  Day 57 | 30.0 [6.7 to 65.2] | 100.0 [69.2 to 100.0] | 20.0 [2.5 to 55.6] | 100.0 [66.4 to 100.0] | 33.3 [7.5 to 70.1] | 80.0 [44.4 to 97.5]
  Day 64: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 9
  Day 64 | 50.0 [18.7 to 81.3] | 100.0 [69.2 to 100.0] | 40.0 [12.2 to 73.8] | 100.0 [66.4 to 100.0] | 50.0 [15.7 to 84.3] | 77.8 [40.0 to 97.2]
  Day 85 | 50.0 [18.7 to 81.3] | 100.0 [69.2 to 100.0] | 50.0 [18.7 to 81.3] | 100.0 [66.4 to 100.0] | 33.3 [7.5 to 70.1] | 90.0 [55.5 to 99.7]
  Day 113: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9 | 10
  Day 113 | 50.0 [18.7 to 81.3] | 100.0 [69.2 to 100.0] | 55.6 [21.2 to 86.3] | 100.0 [66.4 to 100.0] | 33.3 [7.5 to 70.1] | 80.0 [44.4 to 97.5]

9. Secondary Outcome: Peak Fold Rise From Baseline in C. Jejuni Capsule-specific Immunoglobulin G (IgG) Serum Antibody Titer
Description: Serum from blood collected at Study Days 1, 8, 29, 36, 57, 64, 85, and 113 was analyzed using an enzyme-linked immunosorbent assay (ELISA) to measure C. jejuni capsule-specific Immunoglobulin G (IgG) serum antibody titers. Results below the lower limit of quantification (LLOQ) were imputed as LLOQ/2. For each participant, peak fold-rise from baseline is defined as the maximum fold-rise in antibody titer that occurred throughout all follow-up visits with available data (Day 8 up to Day 113) as compared to baseline (Day 1). The peak fold-rise from baseline per participant is summarized by study arm via geometric mean and 95% confidence interval based on Student's t distribution.
Time Frame: Day 8 through Day 113
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise from baseline
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 10
fold rise from baseline | 7.13 [3.27 to 15.53] | 1621.88 [441.35 to 5960.04] | 6.81 [2.13 to 21.82] | 369.59 [163.72 to 834.33] | 5.72 [2.21 to 14.85] | 61.66 [11.96 to 317.83]

10. Secondary Outcome: Maximum C. Jejuni Capsule-specific Immunoglobulin G (IgG) Serum Antibody Titer
Description: Serum from blood collected at Study Days 1, 8, 29, 36, 57, 64, 85, and 113 was analyzed using an enzyme-linked immunosorbent assay (ELISA) to measure C. jejuni capsule-specific Immunoglobulin G (IgG) serum antibody titers. Results below the lower limit of quantification (LLOQ) were imputed as LLOQ/2. For each participant, the maximum antibody titer measured throughout all follow-up visits with available data (Day 8 up to Day 113) was recorded. The maximum post-baseline titer per participant is summarized by study arm via geometric mean and 95% confidence interval based on Student's t distribution.
Time Frame: Day 8 through Day 113
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 10
titer | 1004.6 [518.0 to 1948.4] | 233346.5 [53306.1 to 1021471.1] | 977.2 [305.2 to 3129.1] | 44213.8 [20874.7 to 93647.4] | 812.8 [355.3 to 1859.0] | 9727.4 [2047.9 to 46205.9]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events (AEs) were collected from first study vaccination through the end of study participation (up to Day 420). Solicited AEs and clinical safety laboratory AEs were collected after each study vaccination through 7 days post-vaccination.
Arm/Group | 1 µg CJCV2 | 1 µg CJCV2 + ALFQ | 3 µg CJCV2 | 3 µg CJCV2 + ALFQ | 10 µg CJCV2 | 10 µg CJCV2 + ALFQ
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/10 | 0/9 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 9/10 | 10/10 | 9/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 µg CJCV2 (N=10) | 1 µg CJCV2 + ALFQ (N=10) | 3 µg CJCV2 (N=10) | 3 µg CJCV2 + ALFQ (N=10) | 10 µg CJCV2 (N=9) | 10 µg CJCV2 + ALFQ (N=10)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 µg CJCV2 (N=10) | 1 µg CJCV2 + ALFQ (N=10) | 3 µg CJCV2 (N=10) | 3 µg CJCV2 + ALFQ (N=10) | 10 µg CJCV2 (N=9) | 10 µg CJCV2 + ALFQ (N=10)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heterogeneously dense breasts (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (3) | 1 (1) | 5 (9) | 2 (5) | 5 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (10) | 9 (23) | 4 (8) | 9 (18) | 4 (4) | 8 (17)
Injection site erythema (General disorders) | 2 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 5 (9)
Injection site haemorrhage (General disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 1 (2)
Injection site induration (General disorders) | 0 (0) | 3 (4) | 2 (2) | 4 (6) | 2 (4) | 4 (6)
Injection site pain (General disorders) | 5 (8) | 10 (39) | 5 (8) | 10 (41) | 7 (13) | 9 (37)
Malaise (General disorders) | 5 (7) | 9 (18) | 2 (3) | 8 (15) | 5 (6) | 9 (15)
Pyrexia (General disorders) | 0 (0) | 6 (11) | 0 (0) | 6 (12) | 1 (1) | 7 (11)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (4) | 1 (1) | 2 (3) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 2 (2) | 3 (4) | 3 (5) | 3 (5) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (9) | 0 (0) | 4 (5) | 1 (1) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 10 (25) | 3 (3) | 9 (19) | 2 (3) | 8 (16)
Headache (Nervous system disorders) | 6 (9) | 10 (19) | 5 (7) | 7 (18) | 6 (8) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT05500417/Prot_001.pdf
  • Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT05500417/SAP_002.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT05500417/ICF_000.pdf